CLINICAL TRIAL: NCT04032288
Title: Establish a Prospective Registration System of ARDS Patients for Improving Quality of Care
Status: Completed | Type: Observational
Sponsor: Chimei Medical Center (Other)
Responsible Party: Principal Investigator, Kuo-Chen Cheng, Consultant, Chimei Medical Center
Other Study IDs: CMFHR10154(IRB10110-009)
Record Dates: First submitted 2018-01-24; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Mortality
Keywords: ARDS; Low tidal volume ventilation; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The registration system will enroll and follow up ARDS patients prospectively through screening patients with bilateral radiographic infiltrates and a PaO2/FiO2 ratio of 200 mmHg or less by respiratory therapist. The diagnosis of ARDS must be made by an intensivist or chest physician. Including characteristics, co-morbidities, clinical features, laboratory data, organs dysfunction, treatments and outcomes of ARDS patients will be recorded.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) is defined as a syndrome of acute and persistent lung inflammation with increased vascular permeability and characterized by three clinical features: bilateral radiographic infiltrates; a PaO2/FiO2 ratio of 200 mmHg or less, regardless of the level of PEEP and no clinical evidence for an elevated left atrial pressure. If measured, the pulmonary capillary wedge pressure is 18 mmHg or less. In 1994, the American-European Consensus Conference on acute respiratory distress syndrome (ARDS) issued the above definitions that have been widely used by clinicians and researchers (1, 2) When patients with acute respiratory distress syndrome (ARDS), an age-adjusted incidence of 64 per 100,000 person-years and a mortality of 41 percent were detected. Within intensive care units, approximately ten to 15 percent of admitted patients and up to 20 percent of mechanically ventilated patients meet criteria for ARDS (3-6). The mortality rate varies on the basis of the underlying cause, with most patients dying of multi-organ system failure rather than isolated respiratory insufficiency (5, 7). Large trials suggest that the overall mortality of ARDS ranges from 26 to 58 percent (8, 9). The better outcomes always came from tertiary medical centers or big clinical trials, which somewhat might conceal the fact of presence of higher mortality. The mortality rate in our hospital ever reached or even up to 67.2%(10). To improve the quality of care in ARDS patients still has a long way to. We hope to establish a prospective registration system to understand the real status of quality of care first, and then quality improvement interventions will be followed.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patients prospectively through screening patients with bilateral radiographic infiltrates and a PaO2/FiO2 ratio of 200 mmHg or less by respiratory therapist.

Exclusion Criteria:

* NA.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARDS patients prospectively through screening patients with bilateral radiographic infiltrates and a PaO2/FiO2 ratio of 200 mmHg or less by respiratory therapist.
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-10-11; Primary Completion 2015-07 (Actual); Study Completion 2016-08-11 (Actual)

PRIMARY OUTCOMES:
mortality | 1 year
  Hospital Mortality Rate

CONTACTS AND LOCATIONS:
Overall Officials: Kuo-Chen Cheng, Chief, Study Chair — Chi Mei Medical Hospital
Locations (1):
- Department of Intensive Care Medicine; Chi Mei Medical Center, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No